CLINICAL TRIAL: NCT00160797
Title: MIS™ Minimally Invasive Solutions™ Total Knee Arthroplasty Outcome Study #02-800
Brief Title: Total Knee Arthroplasty Outcome Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: 10/2005 PI assigned duties as trauma physician in addition other duties
Sponsor: University of Florida (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 580-2004
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Total Knee Replacement

INTERVENTIONS:
Device: MIS™ Minimally Invasive Solutions™ TKA System

SUMMARY:
The purpose of this study is to gather information about total knee replacement surgery using minimally invasive surgical procedures.

DETAILED DESCRIPTION:
The purpose of this study is to gather information about total knee replacement surgery using minimally invasive surgical procedures. The MIS™ Minimally Invasive Solutions™ Total Knee Arthroplasty System has been cleared for use by the Food and Drug Administration.

You are invited to participate in this data collection study, comparing the MIS system to standard knee replacement systems. The decision about which system and operation will be best for you has already been made by you and your orthopaedic surgeon.

The information will be used to compare minimally invasive surgery and the standard surgery procedures. The results of this study will provide information that will add to the knowledge base of knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a severely disabled joint secondary to painful osteoarthritis, rheumatoid arthritis, or post-traumatic arthritis that warrants primary knee arthroplasty.
* Gender - Males and females will be included. The male-to-female ratio will depend upon the patient population at each institution conducting the study.
* Age - Minimum of 18 years-old.
* Stable Health - The patient should be able to undergo surgery and participate in a follow-up program based upon physical examination and medical history.
* Patient or patient's legal representative has read and signed the Letter to the Patient form.

Exclusion Criteria:

* Patient is skeletally immature.
* Previous ipsilateral knee arthroplasty.
* Previous Patellectomy.
* Patient is pregnant or breastfeeding.
* Presence of clinically significant disease of the cardiovascular, renal, hepatic, hematologic, respiratory, endocrine, neurological, gastrointestinal, genitourinary, immune systems or other medical condition which is not well controlled.
* Patients who have received an investigational drug or device within the last 30 days.
* Patient is unwilling or unable to cooperate in a follow-up program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-08; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard G. Vlasak, M.D., Principal Investigator — University of Florida